CLINICAL TRIAL: NCT05250973
Title: A Phase 2, Multicohort Study of Daratumumab-Based Therapies in Participants With Amyloid Light Chain (AL) Amyloidosis
Brief Title: A Study of Daratumumab-Based Therapies in Participants With Amyloid Light Chain (AL) Amyloidosis
Acronym: AQUARIUS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR109160; 54767414AMY2009 (Other: Janssen Research & Development, LLC); 2021-002639-48 (EudraCT Number); 2023-507069-25-00 (Registry Identifier: EUCT number)
Expanded Access: Available
Record Dates: First submitted 2022-02-11; First posted 2022-02-22 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — daratumumab; Cyclophosphamide; Bortezomib; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Participants of Cohort 1 will be randomized to either Arm A or Arm B of Cohort 1 in a 2:1 ratio. For Cohort 2, participants will be enrolled without randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort1 (Arm A): Daratumumab + Immediate Cyclophosphamide, Bortezomib and Dexamethasone (VCd) (Experimental): Participants with newly diagnosed systemic amyloid light chain (AL) amyloidosis with Mayo Cardiac Stage II and IIIa cardiac involvement will receive daratumumab 1800 milligrams (mg) subcutaneously (SC) starting on Day 1 once weekly (q1w) up to Day 22 for cycles 1-2, on Days 1 and 15 for cycles 3-6, and on Day 1 for cycles 7-24 of a 28-day cycle. Participants will also receive VCd (cyclophosphamide 300 milligrams per meter square [mg/m^2] either orally or intravenously [IV], bortezomib 1.3 mg/m^2 SC or IV, dexamethasone 40 mg weekly either orally or IV) weekly starting at Cycle 1 Day 1 up to Day 22 in every 28-day cycle for a maximum of 6 cycles (Cycle 6 Day 22).
  Interventions: Drug: Daratumumab; Drug: Cyclophosphamide; Drug: Bortezomib; Drug: Dexamethasone
- Cohort1 (Arm B): Daratumumab + Deferred VCd (Experimental): Participants with newly diagnosed systemic AL amyloidosis with Mayo Cardiac Stage II and IIIa cardiac involvement will receive SC daratumumab 1800mg on Day 1 once weekly (q1w) up to Day 22 for cycles 1-2, on Days 1 and 15 for cycles 3-6, and on Day 1 for cycles 7-24 of a 28-day cycle. Participants will also receive VCd (Cyclophosphamide 300 mg/m^2 either orally or IV, Bortezomib 1.3 mg/m^2 SC or IV, Dexamethasone 40 mg weekly either orally or IV) starting at Cycle 4 Day 1, weekly (Days 1, 8, 15, 22) in every 28-day cycle for a maximum of 6 cycles (Cycle 9 Day 22).
  Interventions: Drug: Daratumumab; Drug: Cyclophosphamide; Drug: Bortezomib; Drug: Dexamethasone
- Cohort 2: Daratumumab + VCd (Experimental): Participants with racial and ethnic minorities, including Black or African American participants, with newly diagnosed AL amyloidosis will receive SC injection of daratumumab 1800 mg SC on Day 1 once weekly (q1w) up to Day 22 for cycles 1-2, on Days 1 and 15 for cycles 3-6, and on Day 1 for cycles 7-24 of a 28-day cycle. Participants will also receive VCd (cyclophosphamide 300 milligrams per meter square [mg/m^2] either orally or intravenously [IV], bortezomib 1.3 mg/m^2 SC or IV, dexamethasone 40 mg weekly either orally or IV) weekly starting at Cycle 1 Day 1 up to Day 22 in every 28-day cycle for a maximum of 6 cycles (Cycle 6 Day 22).
  Interventions: Drug: Daratumumab; Drug: Cyclophosphamide; Drug: Bortezomib; Drug: Dexamethasone

INTERVENTIONS:
Drug: Daratumumab — Daratumumab will be administered subcutaneously.
  Other Names: JNJ-54767414
Drug: Cyclophosphamide — Cyclophosphamide will be administered either orally or IV.
Drug: Bortezomib — Bortezomib will be administered by SC injection or IV.
Drug: Dexamethasone — Dexamethasone will be administered orally or IV.

SUMMARY:
The purpose of this study is to characterize cardiac safety of Daratumumab, Cyclophosphamide, Bortezomib, and Dexamethasone (D-VCd) treatment regimens (Arm A: daratumumab + immediate VCd treatment and Arm B: daratumumab + deferred VCd) in newly diagnosed systemic amyloid light chain (AL) amyloidosis with cardiac involvement and to identify potential mitigation strategies for cardiac toxicity (cohort 1); to characterize the pharmacokinetics of subcutaneous (SC) daratumumab, among racial and ethnic minorities, including Black or African American, with newly diagnosed AL amyloidosis treated with D-VCd (cohort 2).

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Cardiac involvement (amyloid light chain [AL] amyloidosis Mayo Cardiac Stage II and Stage IIIa) with or without other organ(s) involved; Cohort 2: One or more organs impacted by systemic AL amyloidosis according to consensus guidelines
* Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0, 1 or 2
* A female participant of childbearing potential must have a negative serum or urine test at screening and within 72 hours of the first dose of study treatment and must agree to further serum or urine pregnancy tests during the study
* A male participant must agree not to donate sperm for the purpose of reproduction during the study and for a minimum of 6 months after receiving the last dose of cyclophosphamide or 100 days after discontinuation of daratumumab, whichever is longer
* Cohort 2 only: self-identified racial and ethnic minorities, including Black or African American
* Measurable disease at screening defined by one of the following:

Difference between iFLC and uninvolved FLC (dFLC) >= 40mg/L per central laboratory Serum involved free light chain (iFLC) >= 40 mg/L with an abnormal kappa:lambda ratio Serum M-protein >= 0.5 g/dL

Exclusion Criteria:

* Prior therapy for systemic AL amyloidosis or multiple myeloma including medications that target cluster of differentiation 38 (CD38), with the exception of 160 milligrams(mg) dexamethasone or equivalent corticosteroid maximum exposure prior to randomization/enrollment
* Previous or current diagnosis of symptomatic multiple myeloma, including the presence of lytic bone disease, plasmacytomas, >=60% plasma cells in the bone marrow, or hypercalcemia related to myeloma.
* Participant received any of the following therapies:

  1. treatment with an investigational drug or used an invasive investigational medical device within 14 days or at least 5 half-lives, whichever is less;
  2. vaccinated with an investigational vaccine (except for COVID-19) live, attenuated or replicating viral vector vaccines less than (<) 4 weeks prior to randomization/enrollment. Participants who are taking strong Cytochrome P450 3A4(CYP3A4) inducers must discontinue their use at least 5 half-lives prior to the first dose of bortezomib
* Stem cell transplantation -Planned stem cell transplant during the first 9 cycles of protocol therapy are excluded. Stem cell collection during the first 9 cycles of protocol therapy is permitted
* Grade 2 sensory or Grade 1 painful peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2027-03-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Cardiac Events of Any Toxicity Grade | Up to 12 months
  Number of participants with cardiac events of any toxicity grade will be reported.
Observed Concentration Immediately Prior to the Next Study Treatment Administration (Ctrough) of Daratumumab | Cycle 3 Day 1 predose (each cycle is of 28 days)
  Ctrough is defined as the observed concentration immediately prior to the next study treatment administration.

SECONDARY OUTCOMES:
Overall Complete Hematologic Response (HemCR) Rate | Up to Cycle 12 or Month 12 (whichever occurs later)
  Overall HemCR rate is defined as percentage of participants who achieve HemCR during or after the study treatment.
HemCR Rate | At 6 months
  HemCR rate at 6 month is defined as percentage of participants who achieve HemCR at 6 month during or after the study treatment.
Very Good Partial Response (VGPR) or Better Rate | Up to Cycle 12 or Month 12 (whichever occurs later)
  Hematologic greater than or equal to (>=) VGPR rate is defined as percentage of participants who achieve hematologic response of VGPR or better.
Time to HemCR or (VGPR or Better) | Up to Cycle 12 or Month 12 (whichever occurs later)
  For participants who achieve HemCR (or >=VGPR), time to HemCR (or >=VGPR) is defined as the time between the date of first study treatment and the first efficacy evaluation at which the participant has met all criteria for hematologic complete response (CR) (or >=VGPR).
Duration of Response (HemCR and VGPR or Better) | Up to Cycle 12 or Month 12 (whichever occurs later)
  For participants who achieve HemCR (or >=VGPR), duration of HemCR (or >=VGPR) is defined as the time between the date of initial documentation of HemCR (or >=VGPR) to the date of first documented evidence of hematologic progressive disease or death, whichever comes first.
Organ Response Rate (OrRR) | Up to Cycle 12 or Month 12 (whichever occurs later)
  Organ response rate is defined as the percentage of participants who achieve organ response in each corresponding organ (kidney, heart, liver).
Overall Survival (OS) | Until Cycle 12 or Month 12 (whichever occurs later)
  OS is measured from the date of first study treatment to the date of the participant's death.
Time to Subsequent Therapy | Up to Cycle 12 or Month 12 (whichever occurs later)
  Time to subsequent therapy for amyloid light chain (AL) amyloidosis is defined as the time from the date of first study treatment to the start date of subsequent AL amyloidosis (non-protocol) treatment.
Number of Participants with Adverse Events (AEs) by Severity | Up to Cycle 12 or Month 12 (whichever occurs later)
  Number of participants with AEs by severity will be reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study.
Serum Concentration of Daratumumab | Up to 3 years
  Serum samples will be analyzed to determine concentrations of daratumumab.
Number of Participants with Antibodies to Daratumumab | Up to Cycle 12 or Month 12 (whichever occurs later)
  Number of participants with antibodies to daratumumab will be reported.
Number of Participants with Antibodies to Recombinant Human Hyaluronidase PH20 Enzyme (rHuPH20) | Up to Cycle 12 or Month 12 (whichever occurs later)
  Number of participants with antibodies to rHuPH20 will be reported.
Change from Baseline in Clinical Signs and Symptoms Score of Cardiac AL Amyloidosis | Up to Cycle 12 or Month 12 (whichever occurs later)
  Change from baseline in clinical signs and symptoms score of cardiac AL amyloidosis will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (46):
- United States (16):
  - City of Hope, Duarte, California
  - Smilow Cancer Hospital/Yale Cancer Center, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute Emory University, Atlanta, Georgia
  - Tufts Medical Center, Boston, Massachusetts
  - Boston University Medical Center, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - Wake Forest University - Baptist Medical Center, Winston-Salem, North Carolina
  - University Hospital of Cleveland, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - UT Southwestern Medical Center, Dallas, Texas
  - VCU Medical Center, Richmond, Virginia
  - University of Washington, Seattle, Washington
- Canada (3):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - University Health Network UHN Princess Margaret Cancer Centre, Toronto, Ontario
- China (5):
  - Peking University First Hospital, Beijing
  - Peking University People's Hospital, Beijing
  - West China Hospital Si Chuan University, Chengdu
  - First affiliated Hospital of Zhejiang University, Hangzhou
  - Ruijin Hospital Shanghai Jiao Tong University, Shanghai
- France (4):
  - CHU de Limoges, Limoges
  - Centre hospitalier Lyon-Sud, Pierre-Bénite
  - CHU De Poitiers, Poitiers
  - CHU Rangueil, Toulouse
- Germany (3):
  - Charite Campus Benjamin Franklin, Berlin
  - Universitatsklinikum Essen, Essen
  - Universitaetsklinikum Heidelberg Medizinische Klinik V, Heidelberg
- Alexandra General Hospital of Athens, Athens, Greece
- Italy (3):
  - Università Degli Studi Di Napoli Federico Ii, Napoli
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - DIPARTIMENTO DI BIOTECNOLOGIE CELLULARI ED EMATOLOGIA - UNIVERSITà ''LA SAPIENZA'', Roma
- Netherlands (3):
  - University Medical Center Groningen, Groningen
  - Hospital Maastricht University Medical Center, Maastricht
  - UMC Utrecht, Utrecht
- Spain (6):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp Clinic de Barcelona, Barcelona
  - Clinica Univ. de Navarra, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp Clinico Univ de Salamanca, Salamanca
- United Kingdom (2):
  - Leicester Royal Infirmary - Haematology, Leicester
  - University College Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency